CLINICAL TRIAL: NCT00289029
Title: Visipaque and Isovue in Cardiac Angiography in Renally Impaired Patients
Brief Title: A Study of Two Iodinated Contrast Agents in Renally Impaired Patients Undergoing Cardiac Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IOP104
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: CIN

INTERVENTIONS:
Drug: Iopamidol 370 mgI/mL

SUMMARY:
The main purpose of this study is to compare the incidence of contrast induced nephrotoxicity following the administration of Isovue or Visipaque in patients with moderate to severe renal insufficiency undergoing cardiac angiography. Serum creatinine will be measured before and up to 48-72 hours after the administration of the contrast agent to evaluate renal function.

ELIGIBILITY:
Inclusion Criteria:

* Referred for cardiac angiography; with a documented predose eGFR of greater than or equal to 20 and less than 60 mL/min/1.73m2

Exclusion Criteria:

* Unstable renal function; concurrent administration of nephrotoxic drugs, undergoing dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-07; Study Completion 2006-06

PRIMARY OUTCOMES:
Increase in SCr at 48-72 hours post dose

SECONDARY OUTCOMES:
Decrease in eGFR at 48-72 hours post dose; occurrence of adverse events; effect on heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Marie Morris, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Inc, Princeton, New Jersey, United States